CLINICAL TRIAL: NCT00077415
Title: A Randomized Phase II Study Of Triapine® Alone Versus Triapine and Gemcitabine As Second-Line Treatment Of Advanced Non-Small-Cell-Lung Cancer In Patients Who Had Prior Gemcitabine With Evaluation Of The Effect Of Triapine® On Gemcitabine Pharmacokinetics and Cellular Uptake In Peripheral Mononuclear Cells
Brief Title: 3-AP and Gemcitabine as Second-Line Therapy in Treating Patients With Stage III or Stage IV Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Therapeutics Research Group (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CTRG-LUN012; CDR0000350313 (Registry Identifier: PDQ (Physician Data Query)); NCI-6256
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2006-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Gemcitabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 3-AP and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving 3-AP together with gemcitabine as second-line therapy works in treating patients with recurrent stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with stage III or IV recurrent non-small cell lung cancer treated with 3-AP (Triapine®) and gemcitabine as second-line therapy.

Secondary

* Determine the response duration, median time to progression, and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the effect of 3-AP (Triapine®) on gemcitabine pharmacokinetics and cellular uptake into peripheral mononuclear cells in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to participating center.

Patients receive 3-AP (Triapine®) IV over 4 hours and gemcitabine IV over 30 minutes on days 1, 8, and 15*. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *For course 1 only, gemcitabine is administered alone on day 1 and in combination with 3-AP (Triapine®) on days 8 and 15.

Patients are followed every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 15-31 patients will be accrued for this study within 7.5-21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed* non-small cell lung cancer (NSCLC)

  * Stage III or IV disease
  * One of the following cellular types:

    * Adenocarcinoma
    * Non-diffuse bronchoalveolar cell carcinoma
    * Large cell carcinoma
    * Squamous cell carcinoma NOTE: *A repeat biopsy of any accessible tumor site is required if > 5 years have elapsed since the initial diagnosis
* Progressive disease after 1 prior gemcitabine-containing chemotherapy regimen for stage III or IV NSCLC and must have achieved, at least once, a partial response, complete response, or stable disease during therapy

  * Not a primary non-responder and experienced only progressive disease during gemcitabine-containing chemotherapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No glucose-6-phosphate dehydrogenase (G6PD) deficiency

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No prior uncontrolled cardiac disease
* No myocardial infarction within the past 12 months
* No symptomatic congestive heart failure
* No coronary artery disease
* No cardiac arrhythmia

Pulmonary

* No uncontrolled symptomatic pulmonary disease
* No pulmonary disease that requires oxygen therapy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except completely treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study agents
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2004-04; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Objective tumor response as assessed by RECIST criteria

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0
Overall survival
Median time to progression
Duration of overall response
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, MD, Study Chair — Prince of Wales Hospital
Locations (8):
- Australia (2):
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Singapore (4):
  - Cancer Institute at National University Hospital, Singapore
  - National University of Singapore, Singapore
  - National Cancer Centre - Singapore, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea